CLINICAL TRIAL: NCT07081503
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled Study to Assess ADX-626 in Healthy Participants
Brief Title: Phase 1 Study of ADX-626 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADX-626-101
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADX-626 (Experimental)
  Interventions: Drug: ADX-626
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-626 — siRNA duplex oligonucleotide
  Arms: ADX-626
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
This first-in-human study will evaluate the safety and tolerability of ADX-626 in healthy participants. The study will also look at how ADX-626 interacts with the human body (the pharmacokinetics and pharmacodynamics of ADX-626).

DETAILED DESCRIPTION:
A Phase 1, first-in-human study to assess the safety and tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of ADX-626 compared with placebo in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 to 45 years at the time of informed consent
* Males or women of non-childbearing potential (WONCBP)
* Willing to comply with all study requirements while participating
* Suitable venous access for blood sampling.
* Body weight ≥ 50 kg and a body mass index (BMI) ≤25 kg/m2
* Normal laboratory results including liver enzymes, hemoglobin, platelet count, and coagulation parameters
* Willing to use acceptable contraception methods if applicable

Key Exclusion Criteria:

* Significant medical condition such as hypertension, diabetes, cardiovascular disease, or cancer
* History of bleeding or coagulation disorders, prior instances of major bleeding, or a family history of bleeding disorders.
* Current infection
* Participation in an interventional drug study within the last 90 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Safety of ADX-626 in Healthy Participants | Day 1 to Day 365
  Incidence, relationship and severity of adverse events and serious adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ADX-626 - Maximum Concentration | Day 1 to Day 29
  Cmax
Pharmacokinetics (PK) of ADX-626 - Time to Maximum Concentration | Day 1 to Day 29
  Tmax
Pharmacokinetics (PK) of ADX-626 - Exposure | Day 1 to Day 29
  Area Under the Curve (AUC)
Pharmacodynamics (PD) of ADX-626 - Factor XI | Day 1 to Day 365
  Change from baseline in Factor XI measurements
Pharmacodynamics (PD) of ADX-626 - Blood Clotting Time | Day 1 to Day 365
  Change from baseline in Activated Partial Thromboplastin Time (aPTT)

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Patel, MD, Study Director — ADARx Pharmaceuticals
Locations (1):
- Richmond Pharmacology, London, United Kingdom